CLINICAL TRIAL: NCT03971370
Title: Immunogenicity and Safety of A Lyophilized Purified Human Diploid Cell Rabies Vaccine in Chinese Healthy People Aged 10-60 Years.: A Randomized, Blinded, Phase III Clinical Trial.
Brief Title: Immunogenicity and Safety of A Lyophilized Purified Human Diploid Cell Rabies Vaccine .
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: JSVCT041
Record Dates: First submitted 2019-05-30; First posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Adverse Effect and Immunogenicity of Vaccine
MeSH Terms: interventions — Rabies Vaccines; Long-Term Synaptic Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental 1 (Experimental)
  Interventions: Biological: Human diploid cell rabies vaccine (Minhai Biothechnology Co., Ltd)
- Experimental 2 (Experimental)
  Interventions: Biological: Human diploid cell rabies vaccine (Minhai Biothechnology Co., Ltd)
- Positive Control (Active Comparator)
  Interventions: Biological: Human diploid cell rabies vaccine (Chengdu Kanghua Biological Products Co., Ltd.)

INTERVENTIONS:
Biological: Human diploid cell rabies vaccine (Minhai Biothechnology Co., Ltd) — Essen post-exposure immunization schedule at day 0,3,7,14,28.
  Arms: Experimental 1
Biological: Human diploid cell rabies vaccine (Minhai Biothechnology Co., Ltd) — Zagreb post-exposure immunization schedule at day 0,7,21.
  Arms: Experimental 2
Biological: Human diploid cell rabies vaccine (Chengdu Kanghua Biological Products Co., Ltd.) — Essen post-exposure immunization schedule at day 0,3,7,14,28.
  Arms: Positive Control

SUMMARY:
Rabies is caused by rabies virus with a 100% mortality rate in humans. Most of cases occur in Africa and Asia, mainly in underserved populations. Rabies is a vaccine-preventable disease in both humans and animals. The WHO clearly states that human diploid cell rabies vaccine is the "gold standard" rabies vaccine, because of no carcinogenicity and any foreign animal impurity or neurotoxicity factor. China does not approve the import of foreign HDCV and has insufficiency domestic HDCV, so this clinic trial was to assess the immunogenicity and safety of HDCV in healthy population for the large-scale developing of a lyophilized and purified HDCV.

DETAILED DESCRIPTION:
Rabies is caused by rabies virus with a 100% mortality rate in humans. An estimated 59000 human deaths and over 3.7 million disability-adjusted life years lost every year. Most of cases occur in Africa and Asia, mainly in underserved populations, with approximately 40% of cases in children aged <15 years. WHO and its partners have endorsed a target of Zero Human Rabies Deaths from dog-transmitted rabies by 2030 (Zero by 30). Fortunately, rabies is a vaccine-preventable disease in both humansand animals.

At present, chicken embryo cell vaccine, Vero cell vaccine, hamster kidney cell vaccine, and human diploid cell (HDC) rabies vaccine (HDCV) have been approved. The WHO clearly states that HDCV is the "gold standard" rabies vaccine. Because HDCs are normal karyotype cells without carcinogenicity, the HDCV does not contain any foreign animal impurity or neurotoxicity factor. Furthermore, there are fewer injections required and mild adverse reactions and it is safe and efficacious; thus, it is recommended by the WHO as the "nearly ideal human vaccine." Although HDCV was primarily used in developed countries prior to 2015, China does not approve the import of foreign HDCV. Meanwhile, domestic diploid rabies vaccine for human use is insufficiency and in this regard, Minhai Biothechnology Co., Ltd in China has overcome technical difficulties for the large-scale developing of a lyophilized and purified HDCV. This clinic trial was to assess the immunogenicity and safety of HDCV in healthy population vaccinated according to the Essen and Zagreb post-exposure immunization schedule, exploring the appropriate immunization procedures.

ELIGIBILITY:
Inclusion Criteria:

* - Healthy subjects aged 10-60 years as established by medical history and clinical examination
* The subjects are able to understand and sign the informed consent
* Subjects who can and will comply with the requirements of the protocol
* Subjects with temperature ≤37.0°C on axillary setting

Exclusion Criteria:

* - Subject who was administered human rabies vaccine.
* Suspected or have a history of injury caused by warm-blooded mammals.
* Women who are breastfeeding, pregnant, or planning to become pregnant during the trial.
* Subject that has a medical history of any of the following: allergic history, or allergic to any ingredient of vaccine, especially allergic to neomycin.
* Has been diagnosed or suspected of having an immune deficiency, autoimmune disease, or immune system disorder.
* History of thyroidectomy, or thyroid disease requiring treatmentin the past 12 months
* Bleeding disorder diagnosed by a doctor or significant bruising or bleeding difficulties with injections or blood draws
* History of epilepsy, convulsions or convulsions, or a family history of psychosis.
* Absence of spleen, functional absence of spleen, and any circumstances leading to absence of spleen or splenectomy.
* Have a serious chronic illness (such as Down's syndrome, diabetes, sickle cell anemia or neurological disorders, guillain-barre syndrome)
* Known or suspected co-existing diseases included: respiratory disease, acute infection or active period of chronic disease, HIV infection, cardiovascular disease, severe hypertension, malignant tumor treatment, skin disease.
* In the past 6 months, there have been immunosuppressive therapy, cytotoxic therapy, inhaled corticosteroids (excluding corticosteroid spray therapy for allergic rhinitis, and surface corticosteroid therapy for acute non-complicated dermatitis).
* Taking anti-TB prevention or treatment.
* Any prior administration of blood products in last 3 months.
* Any prior administration of other research drugs in last 30 days
* Any prior administration of attenuated live vaccine in last 14 days
* Any prior administration of subunit or inactivated vaccines in last 7 days
* Had fever 3 days before vaccination, Subjects with temperature ≥38.0°C on axillary setting
* Any condition that in the opinion of the investigator, may interfere with the evaluation of study objectives

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1800 (Actual)
Dates: Start 2017-09-10 (Actual); Primary Completion 2018-09-29 (Actual); Study Completion 2019-02-22 (Actual)

PRIMARY OUTCOMES:
To evaluate immunogenicity after the first dose | 14 days following the first dose
  Percentage of participants with rabies virus neutralizing antibody concentration ≥0.5 IU/ml.

SECONDARY OUTCOMES:
Percentage of participants with rabies virus neutralizing antibody concentration ≥0.5 IU/ml after the last dose. | 14 days following the last dost
  Percentage of participants with rabies virus neutralizing antibody concentration ≥0.5 IU/ml after the last dose.
GMC of rabies virus neutralizing antibody | day 7 and 14 post the first dose and day 14 post the last dose
Proportion of subjects reporting of adverse reaction and unsolicited adverse events | from day 0 to day 28 post the last dose
Proportion of subjects with Serious Adverse Events occurring throughout the trial | Day 0 up to month 12

CONTACTS AND LOCATIONS:
Overall Officials: Yuemei Hu, Master, Principal Investigator — Jiangsu Provincial Center for Diseases Control and Prevention
Locations (1):
- Jiangsu Provincial Center for Diseases Control and Prevention, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Li G, Cao S, Xu B, Hu J, Zhang L, Shi L, Zhao D, Li Y, Liu Y, Liang Q, Wu X. Safety, immunogenicity and immune persistence of a lyophilized purified human diploid cells rabies vaccine following rabies PEP regimen Essen and Zagreb: A randomized, blinded controlled phase 3 trial in healthy participants aged 10-60 years old. Vaccine. 2025 Apr 19;53:127082. doi: 10.1016/j.vaccine.2025.127082. Epub 2025 Apr 5. PMID 40188565